CLINICAL TRIAL: NCT03231709
Title: Treatment Preference for Weekly DPP-4 Inhibitors Versus Daily DPP-4 Inhibitors in Patients With Type 2 Diabetes Mellitus
Brief Title: Treatment Preference for Weekly Dipeptidyl Peptidase-4 (DPP-4) Inhibitors Versus Daily DPP-4 Inhibitors in Participants With Type 2 Diabetes Mellitus
Acronym: TRINITY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Trelagliptin-4003; U1111-1197-5821 (Other: WHO); JapicCTI-173662 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin; alogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trelagliptin 100 mg + Alogliptin 25 mg (Experimental): Trelagliptin preceding group (T-A group): Trelagliptin 100 mg, tablets, orally, once a week for 8 weeks, followed by alogliptin, 25 mg, tablets, orally, once a day for 8 weeks.
  Interventions: Drug: Trelagliptin; Drug: Alogliptin
- Alogliptin 25 mg + Trelagliptin 100 mg (Experimental): Alogliptin preceding group (A-T group): Alogliptin, 25 mg, tablets, orally, once a day for 8 weeks, followed by trelagliptin, 100 mg, tablets, orally, once a week for 8 weeks.
  Interventions: Drug: Trelagliptin; Drug: Alogliptin

INTERVENTIONS:
Drug: Trelagliptin — Trelagliptin tablets
Drug: Alogliptin — Alogliptin tablets

SUMMARY:
The purpose of this study is to examine the participant's preference for treatment with once-weekly dosing of DPP-4 inhibitor trelagliptin versus once-daily dosing of DPP-4 inhibitor alogliptin among the participants with type 2 diabetes mellitus who are being treated with once-daily dosing of DPP-4 inhibitor.

DETAILED DESCRIPTION:
The drugs being tested in this study are called Trelagliptin and Alogliptin. This study will look at the participant's preference for treatment with Trelagliptin versus Alogliptin.

The study enrolled 60 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Trelagliptin 100 mg, followed by Alogliptin 25 mg
* Alogliptin 25 mg, followed by Trelagliptin 100 mg All participants will be asked to take one tablet of trelagliptin orally once a week or one tablet of alogliptin orally once a day throughout the study period.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is 16 weeks. Participants will make 3 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have been diagnosed with type 2 diabetes mellitus.
2. Participants who are being treated with any of the following DPP-4 inhibitors for at least 8 weeks prior to the time of informed consent (Week 0).

   * Sitagliptin : 50 mg once daily
   * Alogliptin : 25 mg once daily
   * Linagliptin : 5 mg once daily
   * Teneligliptin : 20 mg once daily
   * Saxagliptin : 5 mg once daily
3. Participants who were judged by the investigators possible to change the treatment from daily dosing of DPP-4 inhibitor shown in Inclusion Criteria 2 to study drug trelagliptin 100 mg or alogliptin 25 mg.
4. Participants whose glycosylated hemoglobin (HbA1c) value measured within 8 weeks prior to the time of informed consent (Week 0) is below 10.0%.
5. Participants who responded to Diabetes Treatment Satisfaction Questionnaire (DTSQ) at the time of informed consent (Week 0).
6. Participants who were judged by the investigators capable to understand the contents of this clinical research and comply with them.
7. Participants who are able to sign and date the Informed Consent Form before any clinical research procedure begins.
8. Participants who are at least 20 years old at the time of giving the consent.
9. Participants who are classified as outpatients.

Exclusion Criteria:

1. Participants who have a history of taking once-weekly dosing of DPP-4 inhibitor (trelagliptin or omarigliptin).
2. Participants who are being treated with drugs other than those for once-daily oral dosing for the purpose of treatment of chronic complication (for example, "BENET® Tablets 75 mg", a therapeutic agent for osteoporosis which is administered once monthly).
3. Participants who are being treated with twice-daily dosing of DPP-4 inhibitor (vildagliptin or anagliptin).
4. Participants who are being treated with anti-diabetic fixed-dose combination pill contained a DPP-4 inhibitor.
5. Participants with moderate or severe renal impairment (for example, participant whose estimated glomerular filtration rate (eGFR) is below 60 mL/min/1.73m^2).
6. Participants for whom blood sugar control by insulin preparations is desired (for example, participants with severe ketosis, diabetic coma or precoma, type 1 diabetes mellitus, severe infection, or serious trauma before or after surgery).
7. Participants who have a history of hypersensitivity or allergy to DPP-4 inhibitor.
8. Participants with serious heart disease, cerebrovascular disorder, or participants with serious disease in the pancreas, blood, etc.
9. Participants with unstable proliferative diabetic retinopathy.
10. Participants with malignant tumor.
11. Participants who are pregnant, breast-feeding, possibly pregnant, or planning to become pregnant.
12. Participants participating in other clinical studies.
13. Participants who have been determined as inappropriate participants by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - OCROM Clinic, Suita, Osaka
  - ToCROM Clinic, Shinjuku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Meguro S, Matsui S, Itoh H. Treatment preference for weekly versus daily DPP-4 inhibitors in patients with type 2 diabetes mellitus: outcomes from the TRINITY trial. Curr Med Res Opin. 2019 Dec;35(12):2071-2078. doi: 10.1080/03007995.2019.1651130. Epub 2019 Aug 22. PMID 31366262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 18 August 2017 to 4 February 2018.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus (DM) were enrolled in 1 of 2 crossover arms: trelagliptin 100 mg then alogliptin 25 mg or alogliptin 25 mg then trelagliptin 100 mg.
Period: Treatment Period 1
Arm/Group | Trelagliptin 100 mg + Alogliptin 25 mg | Alogliptin 25 mg + Trelagliptin 100 mg
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Reason not Specified | 0 | 1
Period: Treatment Period 2
Arm/Group | Trelagliptin 100 mg + Alogliptin 25 mg | Alogliptin 25 mg + Trelagliptin 100 mg
Started | 30 | 29
Completed | 30 | 28
Not Completed | 0 | 1
Not completed — Pretreatment Event/Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants who received either the investigational product or comparator at least once during the study after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trelagliptin 100 mg + Alogliptin 25 mg | Alogliptin 25 mg + Trelagliptin 100 mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.86) | 59.7 (8.73) | 60.1 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 30 | 30 | 60
Height [Mean (Standard Deviation); unit: cm] | 169.2 (7.44) | 169.9 (6.58) | 169.5 (6.97)
Weight [Mean (Standard Deviation); unit: kg] | 70.57 (10.79) | 69.87 (10.79) | 70.22 (10.70)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 24.61 (3.22) | 24.19 (3.31) | 24.40 (3.24)
Smoking Habits [Count of Participants; unit: Participants]
  Had Smoking Habits | 3 | 7 | 10
  Had No Smoking Habits | 27 | 23 | 50
Alcohol intake history [Count of Participants; unit: Participants]
  Regular Drinker | 19 | 16 | 35
  Occasional Drinker | 1 | 4 | 5
  Non-Drinker | 10 | 10 | 20
Duration of diabetes mellitus [Count of Participants; unit: Participants] — Mean duration between the first diagnosis of type 2 diabetes mellitus and the start of the study was reported.
  Participants
    3 Years or More | 26 | 29 | 55
    Less than 3 Years | 4 | 1 | 5
Glycosylated Hemoglobin A1c (HbA1c) National Glycohemoglobin Standardization Program (NGSP) [Mean (Standard Deviation); unit: percent] — NGSP is the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound.
  percent | 7.34 (0.63) | 7.41 (0.84) | 7.38 (0.74)
Diabetes Treatment Satisfaction Questionnaire (DTSQ) at the time of informed consent [Mean (Standard Deviation); unit: score on a scale] — DTSQ is a self-reported instrument consists of 6 questions about treatment satisfaction and 2 questions regarding blood sugar level. Reported data were calculated by questions excluding Questions 2 and 3, two questions regarding blood sugar level. Each question answered on a 7-point Likert scale from 0 to 6, based on concern with the diabetes treatment and experiences in the past few weeks. Higher total score for questions about treatment satisfaction indicate greater satisfaction with treatment and experiences.
  score on a scale | 23.7 (5.86) | 23.0 (5.48) | 23.3 (5.64)
Work status [Count of Participants; unit: Participants]
  Worker | 24 | 23 | 47
  Unemployed | 6 | 7 | 13
Presence of Cohabiter [Count of Participants; unit: Participants]
  Living alone | 4 | 4 | 8
  Living together | 26 | 26 | 52
Experience in Educational Hospitalization on Diabetes [Count of Participants; unit: Participants]
  Had Experience | 3 | 2 | 5
  Had No Experience | 27 | 28 | 55
Compliance With DPP-4 Inhibitors During 4-Week Before Start of Treatment [Count of Participants; unit: Participants]
  90 Percent or More | 30 | 30 | 60
Number of Oral Drugs/Day at the Start of the Treatment Period, Excluding Study Drug [Count of Participants; unit: Participants]
  1 or 2 Tablet(s) | 12 | 9 | 21
  3 - 5 Tablets | 13 | 11 | 24
  6 Tablets or More | 5 | 10 | 15
Complication of Metabolic Syndrome [Count of Participants; unit: Participants]
  Had Presence of Complications | 11 | 11 | 22
  Had No Presence of Complications | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Their Treatment Preference Using Standardized Questions at the End of Treatment Period
Description: Participants answered standardized questions about their preference of drug therapy for Type 2 Diabetes Mellitus. Participants selected one choice from the following 4 choices; either once-weekly DPP-4 inhibitor or daily DPP-4 inhibitor, once-weekly DPP-4 inhibitor, daily DPP-4 inhibitor, neither once-weekly DPP-4 inhibitor nor daily DPP-4 inhibitor. Reported data was the number of participants with a choice of either trelagliptin (once-weekly DPP-4 inhibitor) or alogliptin (once-daily DPP-4 inhibitor), trelagliptin, alogliptin, neither trelagliptin nor alogliptin.
Time Frame: At Week 16
Population: FAS included all enrolled participants who received either the investigational product or comparator at least once during the study after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 100 mg + Alogliptin 25 mg | Alogliptin 25 mg + Trelagliptin 100 mg
Number analyzed (Participants) | 30 | 30
Participants
  Either Trelagliptin or Alogliptin | 4 | 7
  Trelagliptin | 8 | 10
  Alogliptin | 18 | 13
  Neither Trelagliptin nor Alogliptin | 0 | 0
Statistical Analysis 1: Comparison: Trelagliptin 100 mg + Alogliptin 25 mg vs Alogliptin 25 mg + Trelagliptin 100 mg; Test type: Other; p = 0.0141, Mainland-Gart Test

2. Secondary Outcome: Number of Participants by Their Treatment Preference Using Standardized Questions at the End of Treatment Period by Background Factors
Description: Participants answered standardized questions about their preference of drug therapy for Type 2 Diabetes Mellitus. The preference of drug therapy was categorized by background factors like age (years), gender, height (cm), weight (kg), BMI (kg/m^2), duration of diabetes (years), work status, alcohol intake history, smoking habits, experience of educational hospitalization on DM, presence of cohabiter, percentage of compliance with DPP-4 inhibitors during 4-weeks before the start of treatment period, number of oral drugs per day at the beginning of treatment period (excluding investigational drug), complication of metabolic syndrome, percentage of HbA1c (NGSP is the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at the time of informed consent.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Either Trelagliptin or Alogliptin: Participants who prefer either trelagliptin 100 mg, tablets, once a week or alogliptin 25 mg, tablets once a day.
- Trelagliptin Preference: Participants who prefer trelagliptin 100 mg, tablets, once a week.
- Alogliptin Preference: Participants who prefer alogliptin 25 mg, tablets, once a day.
- Neither Trelagliptin Nor Alogliptin: Participants who prefer neither trelagliptin 100 mg, tablets, once a week nor alogliptin 25 mg, tablets once a day.
Arm/Group | Either Trelagliptin or Alogliptin | Trelagliptin Preference | Alogliptin Preference | Neither Trelagliptin Nor Alogliptin
Number analyzed (Participants) | 11 | 18 | 31 | 0
Participants
  Age, Min <= - <65 | 9 | 13 | 16 | 0
  Age, 65 <= - <75 | 2 | 5 | 15 | 0
  Gender, Male | 11 | 16 | 27 | 0
  Gender, Female | 0 | 2 | 4 | 0
  Height, Min <= - <150 | 0 | 1 | 0 | 0
  Height, 150 <= - <160 | 0 | 1 | 2 | 0
  Height, 160 <= - <170 | 1 | 9 | 14 | 0
  Height, 170 <= - <=Max | 10 | 7 | 15 | 0
  Weight, Min <= - <50.0 | 0 | 1 | 0 | 0
  Weight, 50.0 <= - <60.0 | 0 | 5 | 5 | 0
  Weight, 60.0<= - <70.0 | 3 | 3 | 12 | 0
  Weight, 70.0 <= - <80.0 | 8 | 6 | 7 | 0
  Weight, 80.0 <= - <=Max | 0 | 3 | 7 | 0
  BMI, Min <= - <18.5 | 0 | 1 | 0 | 0
  BMI, 18.5 <= - <25.0 | 9 | 9 | 18 | 0
  BMI, 25.0 <= - <=Max | 2 | 8 | 13 | 0
  Duration of Diabetes, 3 Years or More | 10 | 17 | 28 | 0
  Duration of Diabetes, Less than 3 Years | 1 | 1 | 3 | 0
  Work Status, Worker | 9 | 16 | 22 | 0
  Work Status, Unemployed | 2 | 2 | 9 | 0
  Alcohol Intake History, Regular Drinker | 5 | 7 | 23 | 0
  Alcohol Intake History, Occasional Drinker | 2 | 3 | 0 | 0
  Alcohol Intake History, Non-Drinker | 4 | 8 | 8 | 0
  Had Smoking Habits | 4 | 4 | 2 | 0
  Had No Smoking Habits | 7 | 14 | 29 | 0
  Had Experience of Educational Hospitalization | 3 | 0 | 2 | 0
  Had No Experience of Educational Hospitalization | 8 | 18 | 29 | 0
  Presence of Cohabiter, Live alone | 1 | 3 | 4 | 0
  Presence of Cohabiter, Living together | 10 | 15 | 27 | 0
  Compliance with DPP-4 Inhibitors, 90% or More | 11 | 18 | 31 | 0
  Number of Oral Drugs per Day, 1 or 2 Tablet(s) | 1 | 7 | 13 | 0
  Number of Oral Drugs per Day, 3 - 5 Tablets | 5 | 8 | 11 | 0
  Number of Oral Drugs per Day, 6 Tablets or More | 5 | 3 | 7 | 0
  Had Complication of Metabolic Syndrome | 4 | 4 | 14 | 0
  Had No Complication of Metabolic Syndrome | 7 | 14 | 17 | 0
  HbA1c (NGSP), < 7.0% | 1 | 6 | 11 | 0
  HbA1c (NGSP), 7.0%<= - <8.0% | 7 | 8 | 14 | 0
  HbA1c (NGSP), 8.0%<= | 3 | 4 | 6 | 0

3. Secondary Outcome: Number of Participants by Their Treatment Preference Using Standardized Questions at the End of Treatment Period by Background Factors (T-A Administered Group)
Description: as for outcome 2
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Either Trelagliptin or Alogliptin | Trelagliptin Preference | Alogliptin Preference | Neither Trelagliptin Nor Alogliptin
Number analyzed (Participants) | 4 | 8 | 18 | 0
Participants
  Age, Min <= - <65 | 4 | 5 | 9 | 0
  Age, 65 <= - <75 | 0 | 3 | 9 | 0
  Gender, Male | 4 | 7 | 15 | 0
  Gender, Female | 0 | 1 | 3 | 0
  Height, Min <= - <150 | 0 | 1 | 0 | 0
  Height, 150 <= - <160 | 0 | 0 | 1 | 0
  Height, 160 <= - <170 | 0 | 3 | 11 | 0
  Height, 170 <= - <=Max | 4 | 4 | 6 | 0
  Weight, Min <= - <50.0 | 0 | 1 | 0 | 0
  Weight, 50.0 <= - <60.0 | 0 | 0 | 4 | 0
  Weight, 60.0<= - <70.0 | 1 | 2 | 5 | 0
  Weight, 70.0 <= - <80.0 | 3 | 4 | 5 | 0
  Weight, 80.0 <= - <=Max | 0 | 1 | 4 | 0
  BMI, 18.5 <= - <25.0 | 4 | 4 | 10 | 0
  BMI, 25.0 <= - <=Max | 0 | 4 | 8 | 0
  Duration of Diabetes, 3 Years or More | 4 | 7 | 15 | 0
  Duration of Diabetes, Less than 3 Years | 0 | 1 | 3 | 0
  Work Status, Worker | 4 | 7 | 13 | 0
  Work Status, Unemployed | 0 | 1 | 5 | 0
  Alcohol Intake History, Regular Drinker | 3 | 4 | 12 | 0
  Alcohol Intake History, Occasional Drinker | 1 | 0 | 0 | 0
  Alcohol Intake History, Non-Drinker | 0 | 4 | 6 | 0
  Had Smoking Habits | 0 | 2 | 1 | 0
  Had No Smoking Habits | 4 | 6 | 17 | 0
  Had Experience of Educational Hospitalization | 2 | 0 | 1 | 0
  Had No Experience of Educational Hospitalization | 2 | 8 | 17 | 0
  Presence of Cohabiter, Live alone | 0 | 2 | 2 | 0
  Presence of Cohabiter, Living together | 4 | 6 | 16 | 0
  Compliance with DPP-4 Inhibitors, 90% or More | 4 | 8 | 18 | 0
  Number of Oral Drugs per Day, 1 or 2 Tablet(s) | 1 | 2 | 9 | 0
  Number of Oral Drugs per Day, 3 - 5 Tablets | 3 | 5 | 5 | 0
  Number of Oral Drugs per Day, 6 Tablets or More | 0 | 1 | 4 | 0
  Had Complication of Metabolic Syndrome | 1 | 1 | 9 | 0
  Had No Complication of Metabolic Syndrome | 3 | 7 | 9 | 0
  HbA1c (NGSP), < 7.0% | 1 | 4 | 3 | 0
  HbA1c (NGSP), 7.0%<= - <8.0% | 1 | 4 | 11 | 0
  HbA1c (NGSP), 8.0%<= | 2 | 0 | 4 | 0

4. Secondary Outcome: Number of Participants by Their Treatment Preference Using Standardized Questions at the End of Treatment Period by Background Factors (A-T Administered Group)
Description: as for outcome 2
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Either Trelagliptin or Alogliptin | Trelagliptin Preference | Alogliptin Preference | Neither Trelagliptin Nor Alogliptin
Number analyzed (Participants) | 7 | 10 | 13 | 0
Participants
  Age, Min <= - <65 | 5 | 8 | 7 | 0
  Age, 65 <= - <75 | 2 | 2 | 6 | 0
  Gender, Male | 7 | 9 | 12 | 0
  Gender, Female | 0 | 1 | 1 | 0
  Height, 150 <= - <160 | 0 | 1 | 1 | 0
  Height, 160 <= - <170 | 1 | 6 | 3 | 0
  Height, 170 <= - <=Max | 6 | 3 | 9 | 0
  Weight, 50.0 <= - <60.0 | 0 | 5 | 1 | 0
  Weight, 60.0<= - <70.0 | 2 | 1 | 7 | 0
  Weight, 70.0 <= - <80.0 | 5 | 2 | 2 | 0
  Weight, 80.0 <= - <=Max | 0 | 2 | 3 | 0
  BMI, Min <= - <18.5 | 0 | 1 | 0 | 0
  BMI, 18.5 <= - <25.0 | 5 | 5 | 8 | 0
  BMI, 25.0 <= - <=Max | 2 | 4 | 5 | 0
  Duration of Diabetes, 3 Years or More | 6 | 10 | 13 | 0
  Duration of Diabetes, Less than 3 Years | 1 | 0 | 0 | 0
  Work Status, Worker | 5 | 9 | 9 | 0
  Work Status, Unemployed | 2 | 1 | 4 | 0
  Alcohol Intake History, Regular Drinker | 2 | 3 | 11 | 0
  Alcohol Intake History, Occasional Drinker | 1 | 3 | 0 | 0
  Alcohol Intake History, Non-Drinker | 4 | 4 | 2 | 0
  Had Smoking Habits | 4 | 2 | 1 | 0
  Had No Smoking Habits | 3 | 8 | 12 | 0
  Had Experience of Educational Hospitalization | 1 | 0 | 1 | 0
  Had No Experience of Educational Hospitalization | 6 | 10 | 12 | 0
  Presence of Cohabiter, Live alone | 1 | 1 | 2 | 0
  Presence of Cohabiter, Living together | 6 | 9 | 11 | 0
  Compliance with DPP-4 Inhibitors, 90% or More | 7 | 10 | 13 | 0
  Number of Oral Drugs per Day, 1 or 2 Tablet(s) | 0 | 5 | 4 | 0
  Number of Oral Drugs per Day, 3 - 5 Tablets | 2 | 3 | 6 | 0
  Number of Oral Drugs per Day, 6 Tablets or More | 5 | 2 | 3 | 0
  Had Complication of Metabolic Syndrome | 3 | 3 | 5 | 0
  Had No Complication of Metabolic Syndrome | 4 | 7 | 8 | 0
  HbA1c (NGSP), < 7.0% | 0 | 2 | 8 | 0
  HbA1c (NGSP), 7.0%<= - <8.0% | 6 | 4 | 3 | 0
  HbA1c (NGSP), 8.0%<= | 1 | 4 | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Trelagliptin 100 mg: Trelagliptin 100 mg tablets, orally, once a week for 8 weeks in either Period 1 or 2.
- Alogliptin 25 mg: Alogliptin 25 mg tablets, orally, once a day for 8 weeks in either Period 1 or 2.
Arm/Group | Trelagliptin 100 mg | Alogliptin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/60
Other Adverse Events (participants affected / at risk) | 4/59 | 1/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 100 mg (N=59) | Alogliptin 25 mg (N=60)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 100 mg (N=59) | Alogliptin 25 mg (N=60)
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT03231709/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT03231709/SAP_001.pdf